CLINICAL TRIAL: NCT04469244
Title: Evaluation of the Use of Radiomics in 18F-FDOPA PET Examinations for the Characterization of Gliomas
Acronym: RADDOPAG
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2020PI063
Record Dates: First submitted 2020-06-25; First posted 2020-07-14 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2020-12

CONDITIONS: Study on the Use of Radiomics in Gliomas of Initial Disgnosis
Keywords: 18F-FDOPA; Glioma; Radiomics
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The evaluation of gliomas in imaging represents a real challenge today, at the initial diagnosis, for therapeutic planning or follow-up treatment of these lesions. There is an urgent need for non-invasive imaging tools to evaluate a glioma throughout its management. At present, the diagnosis of certainty is only obtained through an anatomo-pathological analysis with sampling during an invasive procedure (surgery or biopsy). Magnetic resonance imaging, through perfusion, diffusion imaging or spectroscopy is developing in gliomas. However, it remains time-consuming and is not always available. At the same time, positron emission tomography (PET) with amino acids is an interesting alternative for these brain tumours. Amino acid PET has the advantage of being more specific than the abnormalities detected in MRI and the amino acid radiotracers cross the blood-brain barrier, even if not broken, unlike Gadolinium in MRI. Among these radiotracers, 18F-FDOPA can, among other things, assist in the non-invasive staging of gliomas at initial diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient having performed a PET/CT examination at 18F-FDOPA for his glioma in the nuclear medicine department of the CHRU de Brabois for which the raw data are available;
* Person who received full information on the organization of the research and did not object to the use of these data;
* Patients affiliated to a social security scheme

Exclusion Criteria:

* - Person who received full information on the organization of the research and who objected to the use of the data
* Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice).
* A person of full age who is unable to give consent and who is not subject to a legal protection measure.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: common population that underwent a PET/CT scan at 18F-FDOPA for its glioma
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance (sensitivity, specificity, accuracy) of parameters extracted from radiomic analysis to predict the molecular characteristics of gliomas at initial diagnosis. | 1 year
  Evaluating the performance of radiomics use in gliomas at initial diagnosis

SECONDARY OUTCOMES:
Diagnostic performance (sensitivity, specificity, accuracy) of parameters extracted from radiomic analysis to predict glioma recurrence | 1 year
  Assessing the performance of radiomics use in the search for glioma recurrence
Diagnostic performance (sensitivity, specificity, accuracy) of parameters extracted from radiomic analysis to predict the response to glioma treatments. | 1 year
  Evaluating the performance of the use of radiomics in the follow-up of glioma disease treatments
Comparison of dynamic parameters (time to peak, slope, area under curve) obtained with different reconstruction parameters versus dynamic parameters obtained on digital phantom from literature data | 6 months
  Optimization of dynamic analysis for the interpretation of the PET/CT examination at 18F-FDOPA
Comparison of dynamic parameters (time to peak, slope, area under curve) obtained with different reconstruction parameters versus dynamic parameters obtained on digital phantom from literature data | 1 years
  Comparison of diagnostic performance of radiomics, static and dynamic parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU of Nancy, Vandœuvre-lès-Nancy, France